CLINICAL TRIAL: NCT01981083
Title: Randomized, Open Label, Controlled Clinical Trial of Egg Albumin-Based Protein Supplement Versus Renal Specific Oral Supplement in Hemodialysis Patients
Brief Title: Egg Albumin-Based Protein Supplement Versus Renal-specific Supplement in Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Medico Lic Adolfo Lopez Mate (Other Government)
Responsible Party: Principal Investigator, Rafael Gonzalez-Toledo, Affiliated Physician of the Nephrology Service, Centro Medico Lic Adolfo Lopez Mate
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217B500602013026
Record Dates: First submitted 2013-10-30; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Protein-Energy Malnutrition; Kidney Failure, Chronic; Hemodialysis
Keywords: Protein-Energy Malnutrition; Chronic Kidney Disease; Malnutrition-Inflammation Score; Subjective Global Assessment; Hemodialysis; Egg albumin
MeSH Terms: conditions — Protein-Energy Malnutrition; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Egg albumin-based protein supplement (Experimental): Powder form, dosage 30 g daily, duration 6 months
  Interventions: Dietary Supplement: Egg albumin-based protein supplement
- Renal-specific oral supplement (Active Comparator): Liquid form, dosage 237 ml (one can) daily, duration 6 months
  Interventions: Dietary Supplement: Renal-specific oral supplement

INTERVENTIONS:
Dietary Supplement: Egg albumin-based protein supplement
  Other Names: Pure ProEgg
  Arms: Egg albumin-based protein supplement
Dietary Supplement: Renal-specific oral supplement
  Other Names: Enterex Renal
  Arms: Renal-specific oral supplement

SUMMARY:
Malnutrition is seen frequently in hemodialysis units in most developing countries. Malnutrition increases morbidity and mortality in this population and its treatment improves patient survival and health status The purpose of this study is to compare two strategies to improve nutritional status in hemodialysis patients: renal-specific oral supplement (237 ml) versus egg albumin-based protein supplement (30 g) on a daily basis.

This trial uses the Malnutrition Inflammation Score (MIS) and Subjective Global Assessment (SGA) in addition to most used biochemical markers to determine nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease in Hemodialysis

Exclusion Criteria:

* Infection
* Liver insufficiency
* Cancer or neoplasia
* Acquired immunodeficiency syndrome
* Intestinal malabsorption syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change in Malnutrition-Inflammation Score | Bimonthly, up to six months
Change in Subjective Global Assessment | Bimonthly, up to six months

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Lic. Adolfo López Mateos, Toluca, State of Mexico, Mexico